CLINICAL TRIAL: NCT06594263
Title: Cross-cultural Adaptation and Validation of the French Version of the PAPA (Perinatal Assessment of Paternal Affectivity) Self-questionnaire Assessing the Psychological Experience of Fathers Pre- and Post-natal
Brief Title: Validation of the French Version of the Perinatal Assessment of Paternal Affectivity (PAPA)
Acronym: French-Papa
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 VENDITTELLI 2
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-08

CONDITIONS: Perinatal Depression; Affective Disorder; Fathers
Keywords: Fathers; Perinatal; Cross-cultural adaptation; Validation; Depression; Affective disorders; Screening
MeSH Terms: conditions — Mood Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The transition to parenthood is a critical period for both the woman and her partner, and this can affect the mental health of the parents. Like mothers, fathers are at risk of stress, anxiety, depression and post-traumatic stress disorder during the perinatal period.

Existing screening or diagnostic tools have been developed on the basis of traditional depressive symptoms expressed by women. However, the manifestations of perinatal mental disorders appear to be different in men. It is therefore essential to develop tools that are sensitive and specific to both gender and the perinatal period in order to increase the sensitivity and specificity of screening for fathers.

In France, to the best of the knowledge of the investigators, there is no validated tool in French to assess paternal psychological disorders, either prenatally or postnatally. Baldoni et al. had validated a brief self-report questionnaire, the " Perinatal Assessment of Paternal Affectivity " (PAPA), to screen for perinatal signs and symptoms of paternal affective disorder, using a gender-sensitive approach.

The aim of this study is to cross-cultural adapt the PAPA in French and to evaluate its psychometric properties.

This validation of the French-PAPA would provide a simple tool, easy to use in everyday practice, to detect any signs or symptoms of paternal psychopathological distress in the pre- and postnatal period.

DETAILED DESCRIPTION:
The cross-cultural adaptation of the pre- and postnatal versions of the PAPA in French will be conduct according to international guidelines.

The PAPA consists of 8 items assessing in the last two weeks anxiety, depression, perceived stress, irritability/anger, relationship problems, abnormal illness behavior, physiological problems, and addictions and other risky behaviors. The severity of the symptoms and behaviors is rated on a 4-point Likert scale from 0 (not at all) to 3 (a lot). A total score is calculated by summing the 8 items' scores. Three additional items consist of: perceiving the symptoms as related to fatherhood, feeling happy with being or becoming a father, reporting additional aspects to better describe feelings.

The study will be offered to all eligible couples. Recruitment will take place in two different ways, depending on whether it is prenatal or postnatal. Women in the prenatal period will be included during one of the third trimester pregnancy monitoring consultations or during one of the third trimester ultrasounds or during a third trimester parenthood preparation course. If the woman is alone at the consultation, she will be asked if she can bring her partner to the next consultation. Postnatal enrolment will take place in the maternity unit, after the woman has given birth.

The couple will give written informed consent if they agree to participate in the study. The women will not be asked to complete any questionnaires. Only some of their socio-demographic and medical data, and that of their child, will be collected from their electronic medical file. For the prenatal study period, the male partners will complete the study questionnaires online after the consultation in the third trimester of pregnancy, and before the baby is born. For the postnatal study period, the male partners will complete the study questionnaires online eight weeks after the baby's birth.

To assess the test-retest reliability of the French-PAPA, the male partners will receive an e-mail to complete the French-PAPA questionnaire a second time online 10 days after the first completion.

ELIGIBILITY:
Inclusion Criteria:

* Woman and its male partner aged 18 years old and older
* Couple understanding, speaking and reading French
* Couple giving their informed consent to participate voluntarily

Exclusion Criteria:

* Woman without male partner
* Woman admitted to intensive care after giving birth
* Couple whose newborn died peripartum
* Couple who have had a medical abortion or fetal death in utero for the current pregnancy
* Woman and/or male partner refusing to participate in the study
* Woman and/or male partner not speaking French
* Woman and/or male partner in the incapacity to answer the questionnaires
* Woman and/or male partner under guardianship or conservatorship, deprived of liberty, or in the custody of correctional authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and their male partners whose wives have been consulted during the third trimester of pregnancy at the Clermont-Ferrand University Hospital Centre (France) or at one of the three private practices participating in the study and who wish to give birth at the Clermont-Ferrand University Hospital Centre and/or couples whose wives have given birth at the maternity unit of the Clermont-Ferrand University Hospital Centre.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
French-PAPA | 0 day
  Psychometric properties (acceptability, internal validity, validity of structure against external criteria) of the French version of the PAPA questionnaire
Change of French-PAPA from baseline at 10 days | 0 day, 10 days
  Test-retest reliability of the French version of the PAPA questionnaire

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 0 day
  The HADS is a valid and reliable self-report questionnaire that assesses anxiety and depression symptoms. It consists of 14 items, 7 for the anxiety subscale and 7 for the depression subscale. A total score ranging from 0 to 21 is calculated for both subscales, with higher scores representing a higher level of symptoms.
Perceived Stress Scale - 10 items (PSS-10) | 0 day
  The PPS-10 is a widely used self-report questionnaire that evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month. It consists of 10 items rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). A total score is calculated by reverse-scoring questions 4, 5, 7 and 8 and then adding scores of all 10 items together. The total score range from 0 to 10 with higher scores indicating higher perceived stress.
General Health Questionnaire - 12 items (GHQ-12) | 0 day
  The GHQ-12 is a screening self-report instrument to detect psychiatric disorders in community settings and non-psychiatric clinical settings. The scores typically used for items are the binary scale (0-0-1-1) and the 4-point Likert-type scale (0-1-2-3). Responses to all items are summed up to a total score ranging from 0 to 12 (binary scale) or 0 to 36 (Likert scale), with higher scores indicating more severe impairment.
Dyadic Adjustment Scale - 4 items (DAS-4) | 0 day
  The DAS-4 is a self-report questionnaire consisting of 4 items and measuring relationship quality in married or cohabiting couples. Each item is rated on 6-point Likert scale. A total score is obtained by summing all the item scores and ranges from 0 to 20, with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress.
Socio-demographic and medical characteristics of male partners | 0 day
  Age, educational level, professional status, number of children, experience of miscarriage, death in utero or death within 28 days of birth with a current or former partner, use of toxic substances (tobacco, alcohol, cannabis, other substances), health problems, psychological or psychiatric support (during life, currently), tranquillisers, antidepressants, anxiolytics treatments (during life, currently), problems or conflicts at work in the last 6 months, stressful life events in the last 6 months.
Socio-demographic and medical characteristics of female partners | 0 day
  Age, marital status, educational level, professional status, parity, number of embryos at the start of pregnancy, diseases related to pregnancy, hospitalisation during pregnancy.
  Only for couples included in the postnatal period, data on childbirth and the postnatal period : gestational age at delivery, onset of labor, anaesthesia before and after birth, mode of delivery, length of labor, postpartum hemorrhage, transfer of the mother, postnatal pathology, length of mother's stay in the maternity unit.
  Only for couples included in the postnatal period, data on the newborn: weight, gender, reanimation in the delivery room, neonatal transfer, neonatal pathology, length of newborn's stay in the maternity unit, breastfeeding on discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Vendittelli, PhD, Principal Investigator — Clermont-Ferrand University Hospital Centre
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No